CLINICAL TRIAL: NCT00069563
Title: John F. Kennedy Center for Mental Retardation: Parent Vs. Teacher-Training in Children's Mental Health Services
Brief Title: Improving Mental Health Services for Economically Disadvantaged Children: Training Teachers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2P30HD015052 (NIH); 2P30HD015052 (NIH); 1R01MH054237 (NIH); NICHD-0521
Record Dates: First submitted 2003-09-29; First posted 2003-09-30 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Psychopathology
Keywords: Internalizing psychopathology; Externalizing psychopathology

INTERVENTIONS:
Behavioral: Reaching Educators, Children, and Parents (RECAP)

SUMMARY:
Children from low socioeconomic levels are more likely to have a mental disorder. However, they are less likely to receive appropriate treatment for that disorder than are children at higher socioeconomic levels. This study will evaluate a program designed to improve mental health services for these children through public school systems.

DETAILED DESCRIPTION:
Approximately 12% of children under 18 years of age in the United States suffer from a mental disorder; estimates for socioeconomically disadvantaged children are 20% or higher. Unfortunately, these at-risk children often do not receive the needed mental health services either because of a lack of accessible services or because their families lack the motivation or resources to obtain services. In many instances, it is difficult or impossible to involve parents in their children's services. Increased access to services for socioeconomically disadvantaged children is critical. However, increased access alone is not sufficient to meet this population's mental health needs. Effective services must be provided. This study will increase the accessibility of mental health services by providing them in the children's schools and will determine whether teachers can be effective substitutes for parents as the therapeutic change agent. The study will accomplish these objectives through implementation and evaluation of the Reaching Educators, Children, and Parents (RECAP) program.

The RECAP program involves individual and small group sessions with children, classroom groups with the child's broader peer groups, and instruction for classroom teachers and parents. The specific techniques are selected to target the areas thought to be responsible for perpetuating the children's problems. The child component, for example, focuses on: 1) social skills (e.g., how to resolve conflicts non-aggressively; use of humor to deflect teasing); 2) communication skills; 3) improving self-monitoring and self-control; 4) reattribution training (for both hostile attributions and negative self-attributions); 5) setting short- and long-term goals and relating behavior to long-term goals; and 6) relaxation. The program also focuses on motivational issues and helping children understand what is in their best long-term self-interest.

Children in need of but not currently receiving mental health services will be selected from six schools serving high-risk neighborhoods in the Metro Nashville School System. Children will be chosen based on severity of psychopathology. Children will be randomly assigned to receive either: 1) mental health services containing a parent-training component; 2) mental health services containing a teacher-training component; or 3) a no-services control group. All children and their classroom peers will be assessed for behavioral, emotional, and social functioning.

ELIGIBILITY:
Inclusion Criteria

* Enrolled in the 4th grade in a participating public school
* Elevated levels of internalizing or externalizing psychopathology

Exclusion Criteria

* Psychosis in parent(s) or child
* No legal guardian (e.g., state custody)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93
Dates: Start 1995-09; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: Travis Thompson, Ph.D., Principal Investigator — Vanderbilt University; Bahr Weiss, Ph.D., Study Director — Vanderbilt University
Locations (1):
- Department of Psychology and Human Development, Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Background] Weiss B, Harris V, Catron T, Han SS. Efficacy of the RECAP intervention program for children with concurrent internalizing and externalizing problems. J Consult Clin Psychol. 2003 Apr;71(2):364-74. doi: 10.1037/0022-006x.71.2.364. PMID 12699030